CLINICAL TRIAL: NCT06376266
Title: Aged and Elderly Individuals
Brief Title: Assessment of the Intervention Effectiveness of Branched-chain Amino Acids(BCAA) Combined With Medium-chain Fatty Acid(MCFA) Products in Sarcopenia Among Middle-aged and Elderly Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202305083RSC
Record Dates: First submitted 2024-01-04; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-01

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; branched-chain amino acids(BCAA); medium-chain fatty acid(MCFA)
MeSH Terms: conditions — Sarcopenia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receive a daily supplement of branched-chain amino acids combined with medium-chain triglycerides (Active Comparator): receive a daily supplement of branched-chain amino acids combined with medium-chain triglycerides
  Interventions: Combination Product: nutritional supplements
- receive a daily supplement of maltodextrin of the same packaging and quantity (Placebo Comparator): receive a daily supplement of maltodextrin of the same packaging and quantity
  Interventions: Combination Product: nutritional supplements

INTERVENTIONS:
Combination Product: nutritional supplements — a daily supplement of branched-chain amino acids combined with medium-chain triglycerides

SUMMARY:
Taiwan entered an aging society in 2018 and is expected to transition into a super-aged society by 2025. With the increasing elderly population, age-related diseases pose urgent challenges to modern society. According to the Ministry of Health and Welfare's National Health Statistics in 2018, the prevalence of sarcopenia in Taiwan among individuals aged 65 and older is 23.6% for males and 18.6% for females. Sarcopenia, characterized by the loss of skeletal muscle mass due to aging, coupled with decreased muscle strength and/or reduced physical performance, poses a significant risk for disability, decreased quality of life, and increased mortality.

Existing research indicates that appropriate nutrition and exercise can slow the onset of sarcopenia and even increase muscle mass to reverse its effects. This study is an interventional clinical trial recruiting middle-aged and elderly patients with sarcopenia or pre-sarcopenia. The intervention involves a combination of branched-chain amino acids and medium-chain triglyceride products, and the study aims to assess the effectiveness of this intervention for sarcopenia in middle-aged and elderly individuals.

DETAILED DESCRIPTION:
Project Rationale:

Taiwan entered an aging society in 2018 and is expected to transition into a super-aged society by 2025. With the increasing elderly population, age-related diseases pose urgent challenges to modern society. According to the Ministry of Health and Welfare's National Health Statistics in 2018, the prevalence of sarcopenia in Taiwan among individuals aged 65 and older is 23.6% for males and 18.6% for females. Sarcopenia, characterized by the loss of skeletal muscle mass due to aging, coupled with decreased muscle strength and/or reduced physical performance, poses a significant risk for disability, decreased quality of life, and increased mortality.

Existing research indicates that appropriate nutrition and exercise can slow the onset of sarcopenia and even increase muscle mass to reverse its effects. This study is an interventional clinical trial recruiting middle-aged and elderly patients with sarcopenia or pre-sarcopenia. The intervention involves a combination of branched-chain amino acids and medium-chain triglyceride products, and the study aims to assess the effectiveness of this intervention for sarcopenia in middle-aged and elderly individuals.

Project Objectives:

Evaluate the effectiveness of branched-chain amino acids combined with medium-chain triglyceride products as an intervention for sarcopenia in middle-aged and elderly individuals.

Methods:

The study cohort will be recruited from National Taiwan University Hospital, targeting individuals aged 50 and above with sarcopenia or pre-sarcopenia. Randomized double-blind allocation will divide participants into intervention and control groups, with each group recruiting 40 subjects (80 participants in total). The intervention group will receive a daily supplement of branched-chain amino acids combined with medium-chain triglycerides, while the control group will be given maltodextrin of the same packaging and quantity as a placebo.

The study will assess various physiological parameters and functional fitness items, conducting the same tests after an 8-week period to evaluate the effectiveness of branched-chain amino acids combined with medium-chain triglyceride products for sarcopenia intervention in middle-aged and elderly individuals.

Expected Outcomes:

Confirmation of the efficacy of nutritional supplements primarily consisting of branched-chain amino acids and medium-chain triglycerides in intervening in muscle loss and promoting daily life functionality in middle-aged and elderly individuals.

Enhanced understanding of the etiology, diagnosis, and assessment methods of sarcopenia among participating staff.

The study anticipates no patent or other commercial interests. If there are any research developments, they will be owned by National Taiwan University Hospital, with potential applications such as publishing academic papers or technology transfer in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Diagnosis of sarcopenia or pre-sarcopenia

Exclusion Criteria:

* Lack of willingness to participate
* Complete dependence on activities of daily living
* Diagnosis of cancer
* Physician-determined life expectancy of less than two years
* Deemed incapable of undergoing assessment by a physician or clinical assessor

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
the scale of sarcopenia | Baseline, 8 weeks
  muscle mass: this study utilizes BIA or DXA to measure the ASMI (kg/ht^2)
the scale of sarcopenia | Baseline, 8 weeks
  muscle strength: Use a handgrip dynamometer to measure the dominant hand grip strength (kgw) of the participants. Take the maximum value of three measurements, with a one-minute interval between each measurement.
the scale of sarcopenia | Baseline, 8 weeks
  physical performance: During testing, participants are required to cross their arms across their chests and record the time (seconds) taken to perform five consecutive sit-to-stand movements and their walking speed (m/s) over a distance of 6 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-cheng Chan, Dr, Study Director — Department of Geriatrics and Gerontology, National Taiwan University Hospital
Locations (1):
- Department of Geriatrics and Gerontology, National Taiwan University Hospital, Taipei, Taiwan